CLINICAL TRIAL: NCT00881543
Title: "Effect of Dipeptidyl Peptidase IV Inhibitors on Glycemia, Insulin, Glucagon, C Peptide, Glp 1 and Lipids After Isocaloric Meals With Different Nutritional Composition in Patients With Type 2 Diabetes näive of Treatment"
Brief Title: "Effect of Dipeptidyl Peptidase IV After Diets in näive Type 2 Diabetic Patients"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Nanci Valeis, Colaborator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: USaoPauloGH
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Type 2
Keywords: Sitagliptin; Diets; Diabetes type 2; Näive patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dipeptidyl-Peptidase IV Inhibitors; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): This arm will begin taking the placebo by a month, after a month will be tested the diets (the same caloric amount with different composition on fat, protein and carbohydrates)making curves of insulin, glucagon, C peptide and glp 1 and lipid when diets are tested (three acute tests with diets). After that, the patient will begin the drug by month (Januvia, 100 mg a day)and repeat all the three curves using the prepared diets to compare with the first month.
  Interventions: Drug: Dipeptidyl Peptidase IV inhibitors
- 2 (Active Comparator): Since the beginning they will use the drug. Then will make the three tests and after will stop the drug by 1 month and come back to do the tests. We objective to demonstrate the washout of the drug clinically.
  Interventions: Drug: Dipeptidyl Peptidase IV inhibitors

INTERVENTIONS:
Drug: Dipeptidyl Peptidase IV inhibitors — Dosage 100 mg each day, once a day, 2 months
  Other Names: Januvia (Merck Sharp Dome); Sitagliptin

SUMMARY:
The purpose of this study is to demonstrate the secretion of glucose, insulin, glucagon, C-peptide and lipid profile after isocaloric diets with different nutritional compounds (fat, protein and carbohydrate food) in drug näive tipo 2 patients.

DETAILED DESCRIPTION:
It is well known that there is a progressive deterioration in beta-cell function over time in type 2 diabetes (DM2), as indicated by the UKPDS (United Kingdom Prospective Diabetes Study), regardless of therapy allocation, albeit conventional (mainly diet), insulin, chlorpropamide, glibenclamide or metformin treatment. Moreover, the pancreatic islet function was found to be about 50% of normal at the time of diagnosis, independent of the degree of insulin resistance, with the reduction in function probably commencing 10-12 years prior to diagnosis and aggravated by increasing fasting plasma glucose levels.

Optimal metabolic control, especially early intensive glycemic control, plays a role in the prevention of progressive beta cell dysfunction and possibly destruction of the betacells with worsening of diabetes. Many reports have shown that induction of normoglycemia in DM2 results in both improved beta cell function and insulin resistance.The major therapeutic drawback using native GLP-1 is its very short half-life of less than 2 minutes, following exogenous administration, as previously indicated due in part to the protease DDP-IV a result, preventing the degradation of native GLP-1 by inhibiting the active of the DDP-IV enzyme has emerged as a therapeutic strategy for enhancing endogenous GLP-1 action in vivo.Considering that, sitagliptin is the first FDA and ANVISA authorized dipeptidyl peptidase-IV (DPP-IV) inhibitor for diabetes treatment and considering the lack of data about DPP-IV inhibitor effect over glucose, glucagon, insulin, C -peptide and fats after isocaloric diets with different nutritional composition in drug näive patients with type 2 diabetes, we designed this study.

ELIGIBILITY:
Inclusion Criteria:

* Drug näive patients with T2DM (for the purpose of this study "drug näive" patients are defined as subjects who have never been treated with an oral antidiabetic agent or subjects who have not taken any antidiabetic agent for at least 12 weeks prior to study entry (Visit 1) and if they had never received antidiabetic agents then never for > 3 months at any time in the past).
* Age in the range of 18 - 78 years inclusive.
* Male, non-fertile female or female of childbearing potential using a medically approved birth control method. A non-fertile female is defined as:

  * post menopausal ( 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40mlU/m)
  * 6 weeks post bilateral oophorectomy with or without hysterectomy
  * post hysterectomy
  * or sterilized by tubal ligation.
* Written informed consent to participate in the study.
* Ability to comply with all study requirements.

Exclusion Criteria:

* Pregnant or lactating female
* A history of type 1 diabetes, diabetes that is result of pancreatic injury, or secondary forms of diabetes, e.g., Cushing´s syndrome and acromegaly, acute metabolic diabetic complications such as ketoacidosis or hyperosmolar state (coma) within the past 6 months.
* Evidence of significant diabetic complications, e.g., symptomatic autonomic neuropathy or gastroparesis.
* Acute infections wich may affect blood glucose control within 4 weeks prior to visit 1 and other concurrent medical condition that may interfere with the interpretation of efficacy and safety data during the study.
* Any of the following within the past 6 months:

  * myocardial infarction (MI) (if the visit one ECG reveals patterns consistent with a MI and the date of the event cannot be determined, then the patient can enter the study at the discretion of the investigator and the sponsor)
  * coronary artery bypass surgery or percutaneous coronary intervention, unstable angina or stroke.
* Congestive heart failure (CHF) requiring pharmacological treatment.
* Any of the following EGC abnormalities; "Torsades de points", sustained and clinically relevant ventricular tachycardia or ventricular fibrillation, second degree AV block (Mobitz 1 and 2 ), third degree AV block, prolonged QTc (>500 msec)
* Malignancy including leukemia and lymphoma (not including basal cell skin cancer) within the last 5 years.
* Liver disease such as cirrhosis or chronic active hepatitis.
* Donation of one unit ( 500ml) or more of blood, significant blood loss equaling to at least one unit of blood within the past 2 weeks or a blood transfusion within the past 8 weeks.
* Chronic insulin (>4 weeks of treatment in the absence of an intercurrent illness) within the past 6 month.
* Chronic oral or parenteral corticosteroid treatment ( > 7 consecutive days of treatment) within 8 weeks prior to visit 1.
* Treatment with growth hormone or similar drugs.
* Treatment with class Ia, Ib and Ic or III anti-arrhythmics.
* Patients who have already been in a study of sitagliptin or another DPP 4 inhibitor.
* Use of other investigational drugs at visit 1, or within 30 days or 5 half-lives of visit 1.
* Any of the following significant laboratory abnormalities:

  * ALT, AST greater than 3 times the upper limit of the normal range at visit 1. *clinically significant renal dysfunction as indicated by serum creatinine levels > or equal 1,5mg/dl in males, > or equal 1,4 mg/dl in females, or a history of abnormal creatinine clearance < 60 ml/m2/24h
  * clinically significant TSH values outside of normal range at visit 1
  * clinically significant laboratory abnormalities, confirmed by repeated measurement, other than hyperglycemia, hyperinsulinemia, and glycosuria at visit 1.
  * fasting triglycerides > 700 mg / dl at visit 1.
* History of active substance abuse (including alcohol) within the past 2 years.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
secretion of glucose, insulin, glucagon, C-peptide and lipid profile after isocaloric diets | One month

SECONDARY OUTCOMES:
Washout of dipeptidyl peptidase IV inhibitors after one month without the drug | One month

CONTACTS AND LOCATIONS:
Overall Officials: Cristina S Oliveira, Pos Grad, Principal Investigator — Sao Paulo General Hospital; Bernardo L Wajchenberg, PhD, Study Director — Sao Paulo General Hospital
Locations (1):
- University of São Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] da Silva Schreiber C, Rafacho A, Silverio R, Betti R, Lerario AC, Lotenberg AMP, Rahmann K, de Oliveira CP, Wajchenberg BL, da Luz PL. The effects of macronutrients composition on hormones and substrates during a meal tolerance test in drugnaive and sitagliptin-treated individuals with type 2 diabetes: a randomized crossover study. Arch Endocrinol Metab. 2022 May 13;66(3):312-323. doi: 10.20945/2359-3997000000478. Epub 2022 May 12. PMID 35551683